CLINICAL TRIAL: NCT04380818
Title: Low Dose Anti-inflammatory Radiotherapy for the Treatment of Pneumonia by COVID-19: Multi-central Prospective Study
Brief Title: Low Dose Anti-inflammatory Radiotherapy for the Treatment of Pneumonia by COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo de Investigación Clínica en Oncología Radioterapia (Other)
Collaborators: Hospital Universitario Madrid Sanchinarro (Other); Hospital del Mar (Other); Hospital Universitari Sant Joan de Reus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IPACOVID
Record Dates: First submitted 2020-05-04; First posted 2020-05-08 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Pneumonia, Viral
Keywords: COVID 19; RADIATION; Anti-inflammatory effects
MeSH Terms: conditions — Pneumonia, Viral; COVID-19 | interventions — Radiotherapy; Hydroxychloroquine; lopinavir-ritonavir drug combination; tocilizumab; Azithromycin; Adrenal Cortex Hormones; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): a control group only receive pharmacological treatment
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: Ritonavir/lopinavir; Drug: Tocilizumab Injection [Actemra]; Drug: Azithromycin; Drug: Corticosteroid; Drug: Low molecular weight heparin; Device: Oxygen supply
- Experimental group (Experimental): an experimental group will receive low-dose lung irradiation
  Interventions: Radiation: Low-dose radiotherapy; Drug: Hydroxychloroquine Sulfate; Drug: Ritonavir/lopinavir; Drug: Tocilizumab Injection [Actemra]; Drug: Azithromycin; Drug: Corticosteroid; Drug: Low molecular weight heparin; Device: Oxygen supply

INTERVENTIONS:
Radiation: Low-dose radiotherapy — Bilateral low-dose lung irradiation: 0.5 Gy in a single fraction. Optionally, additional 0.5 Gy fraction 48h later
  Arms: Experimental group
Drug: Hydroxychloroquine Sulfate — 200 mg/12h for 5 days
  Other Names: Dolquine
Drug: Ritonavir/lopinavir — 400/100 mg/12h for 7-10 days
  Other Names: Kaletra
Drug: Tocilizumab Injection [Actemra] — 600 mg/day for 1-2 doses
  Other Names: Actemra
Drug: Azithromycin — 500 mg/24h for 3 days
Drug: Corticosteroid — Corticosteroids (methylprednisolone/dexamethasone/prednisone)
Drug: Low molecular weight heparin — low molecular weight heparin (LMWH) in prophylaxis of venous thromboembolism
Device: Oxygen supply — Oxygen

SUMMARY:
Low radiation doses produce anti-inflammatory effects, which may be useful in the treatment of respiratory complications of COVID-19. This type of treatment is non-invasive and therefore, a priori, it can be used in all types of patients.

Main objective: To evaluate the efficacy of low-dose lung irradiation as an adjunctive treatment in interstitial pneumonia in patients with COVID-19 by improving the PAFI O2 by 20% measured 48h after treatment with respect to the pre baseline measurement. -irradiation.

DETAILED DESCRIPTION:
Study design: This is a prospective multicenter study in 2 phases:

1. Exploratory phase. It will include 10 patients, to assess the feasibility and efficacy of low-dose lung irradiation. If a minimum efficiency of 30% is not achieved, the study will not be continued.
2. Comparative phase in two groups, a control group, which will only receive pharmacological treatment, and an experimental one. It will include 96 patients, the allocation will be 1: 2, that is, 32 in the control arm and 64 in the experimental arm, which will receive low-dose lung irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old
* Moderate to severe COVID-19 pneumonia with fewer than 8 days of symptom onset and currently receiving standard medication for COVID-19 at appropriate doses
* PAFIO2 of less than 300 mmHg or SaFI02 <315 mmHg
* Patients who are not candidates for admission to the Intensive Care Unit due to age, concomitant diseases or general condition.
* One of the following conditions:

  * or IL6 greater than 40
  * or PCR> 100mg / l

    * D-dimer greater than 1500ng / ml
    * Suspected cytokine release syndrome
* Have read the information sheet and signed the informed consent

Exclusion Criteria:

* Age <18 years
* Failure to meet the inclusion criteria
* Leukopenia <1000
* Pregnancy
* Not understanding or refusing the purpose of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-09-04 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of low-dose pulmonary irradiation assessed by change in PAFI O2 by 20% | Day 2 after interventional radiotherapy
  To evaluate the efficacy of low-dose pulmonary irradiation as an adjunctive treatment in interstitial pneumonia in patients with COVID-19 by improving the PAFI O2 by 20% measured 48h after treatment with respect to baseline pre-irradiation measurement. .
  In cases of impossibility the SaFiO2 will be determined

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Day 30 and day 90 after interventional radiotherapy
  Lung toxicity measured according to CTCAEv5
Change of the radiological image | Days 7 and day 30 after interventional radiotherapy
  Chest CT
Overall mortality | Day 15 and Day 30 after interventional radiotherapy
  Death of any cause
Measure of pro-inflammatory interleukins | Days 1, day 4 and day 7 after interventional radiotherapy
  Interleukins IL-6, IL-10, IL-1, IL-2, IL-8 (pg/ml)
Measure of trasforming growth factor (TGF-b) | Days 1, day 4 and day 7 after interventional radiotherapy
  TGF-β (ng/ml)
Measure of tumor necrosis factor alpha (TNF-a) | Days 1, day 4 and day 7 after interventional radiotherapy
  TNF-α (pg/ml)
Determining overexpression of pro-inflammatory selectin | Days 1, day 4 and day 7 after interventional radiotherapy
  Overexpression of L-, E-, and P-selectin
Determining cell adhesion molecules (CAMs) | Days 1, day 4 and day 7 after interventional radiotherapy
  Overexpression of ICAM-1, VCAM
Measure of marker of oxidative stress PON-1 | Days 1, day 4 and day 7 after interventional radiotherapy
  PON-1(paraoxonase and arylesterase activity) (IU/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Angel Montero, MD, PhD, Principal Investigator — Hospital Universitario Madrid Sanchinarro; Manel Algara, MD, PhD, Principal Investigator — Hospital del Mar; Merirxell Arenas, MD, PhD, Principal Investigator — Hospital Universitario Sant Joan de Reus
Locations (3):
- Spain (3):
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - Hospital Del Mar, Barcelona
  - Hospital Universitario Madrid Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Individual epidemiological and clinical data will be shared after recruitment is complete.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Protocol/ICF from approval Individual epidemiological and clinical data after recruitment is complete.

REFERENCES:
- [Background] Conti P, Ronconi G, Caraffa A, Gallenga CE, Ross R, Frydas I, Kritas SK. Induction of pro-inflammatory cytokines (IL-1 and IL-6) and lung inflammation by Coronavirus-19 (COVI-19 or SARS-CoV-2): anti-inflammatory strategies. J Biol Regul Homeost Agents. 2020 March-April,;34(2):327-331. doi: 10.23812/CONTI-E. PMID 32171193
- [Background] Rodel F, Frey B, Manda K, Hildebrandt G, Hehlgans S, Keilholz L, Seegenschmiedt MH, Gaipl US, Rodel C. Immunomodulatory properties and molecular effects in inflammatory diseases of low-dose x-irradiation. Front Oncol. 2012 Sep 25;2:120. doi: 10.3389/fonc.2012.00120. eCollection 2012. PMID 23057008
- [Background] Arenas M, Sabater S, Hernandez V, Rovirosa A, Lara PC, Biete A, Panes J. Anti-inflammatory effects of low-dose radiotherapy. Indications, dose, and radiobiological mechanisms involved. Strahlenther Onkol. 2012 Nov;188(11):975-81. doi: 10.1007/s00066-012-0170-8. Epub 2012 Aug 22. PMID 22907572
- [Background] Arenas M, Gil F, Gironella M, Hernandez V, Biete A, Pique JM, Panes J. Time course of anti-inflammatory effect of low-dose radiotherapy: correlation with TGF-beta(1) expression. Radiother Oncol. 2008 Mar;86(3):399-406. doi: 10.1016/j.radonc.2007.10.032. Epub 2007 Nov 26. PMID 18031855
- [Background] Lodermann B, Wunderlich R, Frey S, Schorn C, Stangl S, Rodel F, Keilholz L, Fietkau R, Gaipl US, Frey B. Low dose ionising radiation leads to a NF-kappaB dependent decreased secretion of active IL-1beta by activated macrophages with a discontinuous dose-dependency. Int J Radiat Biol. 2012 Oct;88(10):727-34. doi: 10.3109/09553002.2012.689464. Epub 2012 May 22. PMID 22545750
- [Background] Calabrese EJ, Dhawan G. How radiotherapy was historically used to treat pneumonia: could it be useful today? Yale J Biol Med. 2013 Dec 13;86(4):555-70. PMID 24348219
- [Background] Calabrese EJ, Dhawan G, Kapoor R, Kozumbo WJ. Radiotherapy treatment of human inflammatory diseases and conditions: Optimal dose. Hum Exp Toxicol. 2019 Aug;38(8):888-898. doi: 10.1177/0960327119846925. Epub 2019 May 6. PMID 31060383
- [Background] Kirkby C, Mackenzie M. Is low dose radiation therapy a potential treatment for COVID-19 pneumonia? Radiother Oncol. 2020 Jun;147:221. doi: 10.1016/j.radonc.2020.04.004. Epub 2020 Apr 6. No abstract available. PMID 32342871
- [Background] Jean-Marc Cosset, Éric Deutsch, Louis Bazire, Jean-Jacques Mazeron, Cyrus Chargari, Irradiation pulmonaire à faible dose pour l'orage de cytokines du covid-19: pourquoi pas?, Cancer/Radiothérapie, 2020, , ISSN 1278-3218, https://doi.org/10.1016/j.canrad.2020.04.003.
- [Background] Dhawan G, Kapoor R, Dhawan R, Singh R, Monga B, Giordano J, Calabrese EJ. Low dose radiation therapy as a potential life saving treatment for COVID-19-induced acute respiratory distress syndrome (ARDS). Radiother Oncol. 2020 Jun;147:212-216. doi: 10.1016/j.radonc.2020.05.002. Epub 2020 May 8. PMID 32437820
- [Derived] Algara M, Arenas M, Marin J, Vallverdu I, Fernandez-Leton P, Villar J, Fabrer G, Rubio C, Montero A. Low dose anti-inflammatory radiotherapy for the treatment of pneumonia by covid-19: A proposal for a multi-centric prospective trial. Clin Transl Radiat Oncol. 2020 Jun 15;24:29-33. doi: 10.1016/j.ctro.2020.06.005. eCollection 2020 Sep. PMID 32613089